CLINICAL TRIAL: NCT00066209
Title: An Investigation of the Inflammatory Response in Severe Acute Respiratory Syndrome (SARS)
Brief Title: Investigating Severe Acute Respiratory Syndrome (SARS)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030240; 03-I-0240
Record Dates: First submitted 2003-08-05; First posted 2003-08-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-05-24

CONDITIONS: SARS Virus
Keywords: Inflammation; Coronavirus; Immunity; Interferon; Cytokine; Severe Acute Respiratory Syndrome; SARS; Healthy Volunteer; HV
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Inflammation; Coronavirus Infections

SUMMARY:
Severe Acute Respiratory Syndrome (SARS) is a newly recognized illness that can be fatal.

The purpose of this study is to better understand SARS by collecting samples of blood and other body fluids of people who have been exposed to SARS or who are suspected to have the illness.

Up to 300 volunteers aged 18 years or older will be enrolled in this study. Participants will donate blood samples and, if appropriate, samples of fluid from the lungs, nose, or throat. Researchers will test these samples for proteins that control or mediate inflammatory or immune responses. The patterns of these proteins will reveal how SARS affects the body and the efforts the body makes to fight off the infection.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome (SARS) is a newly recognized illness associated with substantial mobidity and mortality. Patients develop fever followed by rapidly progressive and even fatal respiratory disease. SARS is associated with infection with a novel coronavirus. The evaluation of the inflammatory responses evoked by SARS may yield information regarding its pathogenesis and help with patient management. This protocol, then, merely aims to study disease pathogenesis and natural history, by studying samples and data that are collected by outside physicians or physicians at the Clinical Center and sent for evaluation of the inflammatory response.

ELIGIBILITY:
* INCLUSION CRITERIA - CASES:

Patients fulfilling the CDC case definition or WHO definition for suspected or probable SARS.

Newly identified patients found to have recovered from SARS can also be enrolled.

EXCLUSION CRITERIA - CASES:

Patients diagnosed with alternative illnesses as the cause of the symptoms.

INCLUSION CRITERIA - HEALTHY VOLUNTEERS:

For the purpose of this study, a healthy volunteer is defined as a healthy male or female, age 18 and above.

Volunteers will be excluded if they have a pre-existing or concurrent serious chronic medical or psychiatric illness.

Chronic medication use will be evaluated on a case-by-case basis.

They will also be excluded if they have received an investigational drug in the past 3 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2003-08-04; Study Completion 2007-05-24

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States